CLINICAL TRIAL: NCT00643630
Title: A Study to Determine the Skin Barrier Effect of Tetrix Cream
Brief Title: Evaluation of Tetrix Cream as a Protective Barrier Against Injurious Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coria Laboratories, Ltd. (Industry)
Responsible Party: D. Innes Cargill, PhD, Coria Laboratories, Ltd.
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 806 805 09 002
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Healthy
Keywords: Tetrix crea; skin barrier; antigen reaction; prevention; The efficacy of Tetrix Cream to prevent an antigen reaction on the skin.

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Twice daily topical application
  Interventions: Device: Tetrix
- 2 (Placebo Comparator): Twice daily topical application
  Interventions: Device: Tetrix

INTERVENTIONS:
Device: Tetrix — Twice daily topical application
  Arms: 1
Device: Tetrix — Twice daily topical application
  Arms: 2

SUMMARY:
To determine if Tetrix Cream,, when applied to the skin, acts as a barrier to prevent injury to the skin

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects who are sensitized to nickel, neomycin, or fragrance mix.

Exclusion Criteria:

* Under 18 years of age.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-10; Primary Completion 2007-10 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Prevention of delayed bype hypersensitivity reaction following application of antigen | up to 96 hours after antigen application

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Fowler, MD, Principal Investigator — Dermatology Specialists
Locations (1):
- Dermatolgoy Specialists, LLC, Louisville, Kentucky, United States